CLINICAL TRIAL: NCT05303597
Title: The Frequency of Superior Cluneal Nerve Entrapment Diagnosed With Ultrasound Guided Nerve Block In Patients With Low Back Pain: A Prospective, Cross-Sectional Study
Brief Title: The Frequency of Superior Cluneal Nerve Entrapment Diagnosed With Ultrasound Guided Nerve Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Busra Sezer Kıral, residency doctor, Istanbul University - Cerrahpasa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IstanbulUC,BSKıral,001
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Low Back Pain; Nerve Entrapment Syndrome; Radiating Pain
MeSH Terms: conditions — Low Back Pain; Charcot-Marie-Tooth Disease; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- diagnostic superior cluneal nerve block (Other): Patients with low back pain will be evaluated by two physicians. The clinical history and physical examination of all patients with low back pain will be taken by the first physician. Patients with a trigger point in the posterior iliac crest will be evaluated by a second physician and diagnostic nerve block will be performed ultrasound-guided with the preliminary diagnosis of superior cluneal nerve entrapment. General Electric LogiqP5 model ultrasound device will be used and lidocaine will be applied between the posterior iliac crest and thoracolumbar fascia, which is viewed under the guidance of ultrasonography, for diagnosis and treatment. Patients who have had a diagnostic injection will be re-evaluated 1 hour later. Patients whose pain is reduced by more than 70% will be diagnosed with superior cluneal nerve entrapment.
  Interventions: Diagnostic Test: ultrasound-guided diagnostic nerve block with lidocaine

INTERVENTIONS:
Diagnostic Test: ultrasound-guided diagnostic nerve block with lidocaine — Patients with a trigger point in the posterior iliac crest will be evaluated by a second physician and diagnostic nerve block will be performed ultrasound-guided with the preliminary diagnosis of superior cluneal nerve entrapment. General Electric LogiqP5 model ultrasound device will be used and lidocaine will be applied between the posterior iliac crest and thoracolumbar fascia, which is viewed under the guidance of ultrasonography, for diagnosis and treatment.

SUMMARY:
Cluneal nerves are a group of pure sensory nerves that provide direct cutaneous innervation to the buttocks. Superior cluneal nerve(SCN) originates from the T11-L5 nerve roots and has at least 3 branches from medial to lateral; these are the medial, intermediate, and lateral branches. Anatomy studies have shown that the medial branch passes 6-7 cm lateral to the midline on the posterior iliac crest. Nerve branches pass through the osteofibrous tunnel formed by the thoracolumbar fascia and the superior edge of the iliac crest, where they can be trapped. Controversial data exist regarding the osteofibrous tunnel. It may not be present in all cases, and in some cases more than one nerve has been shown to pass through the osteofibrous tunnel. As a result, there are discussions about superior cluneal nerve anatomy and there is not enough information.

In patients with superior cluneal nerve entrapment syndrome, low back pain radiates to the upper part of the hip and may cause leg pain that mimics radiculopathy.

The diagnosis is clinical. Diagnostic criteria for superior cluneal nerve (SCN) entrapment; Low back pain involving the iliac crest and buttocks, symptoms aggravated by lumbar movement or posture, trigger point over the posterior iliac crest corresponding to the nerve compression zone, patients report numbness and radiating pain in the SCN area (Tinel sign) when the trigger point is compressed, symptom relief by SCN block at the trigger point.

Prevalence studies of superior cluneal nerve entrapment syndrome are very few. Maigne et al reported superior cluneal nerve entrapment in 1.6% of 1,800 patients with low back pain. Kuniya et al showed that 14% of 834 patients with low back pain met the criteria for superior cluneal nerve entrapment. Superior cluneal nerve entrapment is not as rare as it is thought to be among the causes of low back pain. In Turkey, there is no study showing the prevalence of the superior cluneal nerve or its importance in patients with low back pain.

The aim of this study is to examine the patients who applied to Cerrahpasa Faculty of Medicine, Department of Physical Medicine and Rehabilitation polyclinic with low back pain; To confirm the diagnosis with an ultrasound-guided diagnostic injection test, to determine the importance of superior cluneal nerve entrapment.

DETAILED DESCRIPTION:
Patients with low back pain will be examined by two doctors. The clinical history and physical examination of all patients with low back pain will be taken by the first physician. Patients with a trigger point in the posterior iliac crest will be evaluated by a second physician and diagnostic nerve block will be performed ultrasound-guided with the preliminary diagnosis of superior cluneal nerve entrapment. General Electric LogiqP5 model ultrasound device will be used and lidocaine will be applied between the posterior iliac crest and thoracolumbar fascia, which is viewed under the guidance of ultrasonography, for diagnosis and treatment. Patients who have had a diagnostic injection will be re-evaluated 1 hour later. Patients whose pain is reduced by more than 70% will be diagnosed with superior cluneal nerve entrapment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older with mechanical low back pain for more than 3 months
* Without a history of neurological or psychiatric disease
* No history of inflammatory disease
* Patients without a history of trauma in the last 3 months

Exclusion Criteria:

* Age younger than 18 and over 80
* Having a history of acute trauma in the last 3 months
* Presence of inflammatory rheumatic disease (RA, Ankylosing spondylitis, Polymyalgia rheumatica, vasculitides etc.)
* Patients who have been injected (steroid, hyaluronic acid, etc.) in the last 6 weeks
* Presence of active infection
* The use of anticoagulants that may interfere with the injection
* Presence of bleeding disorder
* Known allergy to injection agents
* Presence of uncontrolled diabetes mellitus and/or hypertension
* Presence of heart failure
* History of malignancy
* Having a history of neurological disease
* Pregnancy, lactation
* Psychiatric disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
More than 70% reduction in pain with diagnostic nerve block | two months
  200 patients who applied to the outpatient clinic with low back pain will be examined and patients with posterior iliac crest pain will be given a diagnostic injection under ultrasound guidance with a preliminary diagnosis of superior cluneal nerve entrapment.

CONTACTS AND LOCATIONS:
Overall Officials: Kenan Akgun, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- İstanbul Üniversitesi - Cerrahpasa (IUC), Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No